CLINICAL TRIAL: NCT02707458
Title: Dose-finding and Proof-of-concept Trial of Probucol to Increase Availability of CSF Apolipoprotein-E
Brief Title: Dosage and Efficacy of Probucol-induced apoE to Negate Cognitive Deterioration
Acronym: DEPEND
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Weston Brain Institute (Other); McGill University (Other)
Responsible Party: Principal Investigator, John C. S. Breitner, Director, Centre for Studies on Prevention of Alzheimer's Disease (StoP-AD), Douglas Mental Health University Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEPEND
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Dementia of the Alzheimer Type; Age-related Cognitive Decline; Mild Cognitive Impairment Due to Alzheimer Disease
Keywords: apolipoprotein E; Alzheimer; pre-clinical; pre-symptomatic; dose-finding; prevention
MeSH Terms: interventions — Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): All subjects will receive probucol, starting with a fixed dose of 600 mg daily following the evening meal. The variable plasma concentrations achieved and the resulting modification in concentration of CSF apoE will suggest an ideal range of plasma concentrations for use of the drug as an inducer of increased availability of apoE in the CSF. The known dose-proportionality of the drug in plasma will then be used to estimate an ideal individualized dose for each participant. The effects of such individualized dosage will be tested over 1 year of follow-up observations, searching for treatment effects on CSF apoE and for evidence of other treatment effects, particularly including adverse effects.
  Interventions: Drug: Probucol

INTERVENTIONS:
Drug: Probucol — Probucol was used with good effect for more than a decade in Canada and the US to reduce plasma cholesterol. Although withdrawn from the Canadian and US markets by its manufacturer for commercial reasons, it is still widely used for this purpose in Japan and Korea. Over the past decade, long-term follow-up studies in Asian populations at high risk of cardiovascular events have shown that the drug reduces the incidence of these events in a manner not unlike "statin" drugs used widely in Canada and the US.
  Other Names: Lorelco (trade name in Japan)

SUMMARY:
DEPEND is an open-label but dosage-masked trial of the retired cholesterol-lowering drug probucol as an agent to increase availability of apolipoprotein E (apoE) in the cerebrospinal fluid (CSF) of cognitively intact older persons at risk of Alzheimer's dementia. Absorption of oral probucol is variable. In a sample of 23 cognitively intact persons over age 55, DEPEND will therefore develop an algorithm to prescribe individualized dosing to achieve plasma concentration that will likely increase availability of CSF apoE. These persons will then use their individualized dosage for 12 months to assess longer-term effects of the drug on CSF apoE concentration, while monitoring closely for evidence of adverse consequences of use.

DETAILED DESCRIPTION:
Probucol is a cholesterol-lowering drug that has been removed from the market in Canada and the US, but remains in clinical use in Asia. In rodents, probucol increases synthesis and availability of apolipoprotein E (apoE) in the cerebrospinal fluid (CSF). ApoE is the protein product of the polymorphic gene APOE, allelic variation in which remains the strongest known risk factor (other than age itself) for Alzheimer's dementia. Oral Probucol is absorbed variably. Administration of a single, fixed dose therefore results in a wide range of plasma concentrations when the drug is given to various individuals in a fixed dosage. Limited human data suggest that higher plasma and CSF concentrations of probucol result in stronger increases in CSF apoE concentration. The dual aims of DEPEND are therefore 1) to develop an individualized dosing regimen that will result in plasma concentrations that are likely to increase CSF apoE concentration by 50%; and 2) to treat 20 persons at elevated risk of Alzheimer's dementia, each at his/her ideal individual dosage, for 12 months, observing the resulting change in CSF concentrations of apoE. Simultaneously, subjects will be observed carefully for evidence of any treatment effects on cognition or other probable markers of progression in pre-clinical Alzheimer's disease, as well as safety risks that might deter further human experimentation with the drug.

ELIGIBILITY:
Inclusion Criteria:

* Family history of one or more parents or multiple siblings who developed Alzheimer-like dementia, as established by review of history and/or medical records, and by responses to a brief questionnaire describing characteristics of the relatives' condition
* Aged 60+. May be aged 55-59 only if at least one parent or sibling experienced onset of Alzheimer's dementia at an age no more than 15 years beyond the prospective participant's current age
* At least six years of formal education
* Sufficient fluency in spoken and written English and/or French to participate in study visits and in psychometric testing
* A collateral respondent available to provide information on the cognitive and health status of the participant, and to assist with monitoring of study interventions, if needed
* Willingness to undergo four lumbar punctures for collection of CSF
* Affirmation of prior informed consent to undergo genetic testing for APOE and other known or suspected AD risk factors
* Ability and intention to participate in study visits per protocol, in the opinion of a study physician
* Willingness to limit use of over-the-counter or prescription medicines (e.g., tricyclic antidepressants, anti-histamines) known to prolong QTc interval, or to potentiate the tendency of probucol to prolong this interval, in the opinion of a study physician
* If on a statin or other lipid lowering drug that, in the opinion of a study physician, can safely be co-administered with probucol, willingness to remain on a stable dose of this medication during the entire trial period.
* Provision of informed consent for this trial.

Exclusion Criteria:

* Known or identified cognitive disorder diagnosed previously by a physician, psychologist, nurse-clinician, or other health care provider, or by StoP-AD staff
* Past or present use of a commercially available acetyl-cholinesterase inhibitor including tacrine, donepezil, rivastigmine, or galantamine
* Past or present use of memantine or other approved cognitive enhancement prescription agent
* History of heart disease, myocardial infarction or documented acute coronary syndrome, or arrhythmia (including atrial fibrillation)
* Corrected QT interval using Bazett's formula (QTcB) interval > 450 msec for males or 470 msec for females as detected by EKG and confirmed by consultant cardiologist
* Clinically significant hypertension, anemia, liver disease, or kidney disease, in opinion of a study physician (participants with treated hypertension who are normotensive as a result of intervention may be enrolled.)
* Concurrent use of over-the-counter or prescription medicines (e.g., tricyclic antidepressants, anti-histamines) known to prolong QTc interval, or to potentiate the tendency of probucol to prolong this interval, in the opinion of a study physician
* Any inflammatory or chronic pain condition that necessitates regular use of opiates (e.g., oxycodone, hydrocodone, tramadol, meperidine, hydromorphone), or NSAIDs (more than 4 doses / week)
* Current plasma creatinine > 132 mmol/l (1.5 mg/dl)
* Current alcohol, barbiturate or benzodiazepine abuse or dependence (in opinion of study physician)
* Any other medical condition that, in the opinion of a study physician, makes it inadvisable for the participant to be assigned to regular dosage of probucol
* Enrolment in any trial or experimental protocol that, in the opinion of a study physician, is likely to interfere with PREVENT-AD or any of its derivative protocols including this one
* Any other condition that, in the opinion of a study physician, makes it medically inappropriate for the participant to enroll in the program

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of probucol following test dose | three months
  Participants are given a test dose of probucol 600 mg q.d. Plasma concentration of probucol and cerebrospinal fluid (CSF) concentrations of probucol and apolipoprotein E (apoE) are measured at baseline and after 3 months. Results should suggest a range of plasma concentrations associated with an increase in CSF apoE by at least 50%. Relying on dose-proportionality of plasma concentration achieved, an estimated optimum individual dose for target levels of apolipoprotein E induction is then calculated.
Apolipoprotein concentration in CSF before and after treatment with probucol at individualized dose | One year on individualized dosing, as suggested by experimental observations above
  After a washout period => 2 months, participants will initiate treatment with probucol at individualized dosage determined in Outcome 1. Results after 1 year will establish whether such individualized dosage of probucol achieves 'target engagement' of specified increase in CSF apoE, to be tested subsequently for its ability to prevent progression of pre-symptomatic Alzheimer disease.

CONTACTS AND LOCATIONS:
Overall Officials: John C Breitner, MD, MPH, Principal Investigator — Douglas Hospital Research Centre & McGill University Faculty of Medicine
Locations (1):
- Douglas Hospital Research Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified data upon completion and publication of trial